CLINICAL TRIAL: NCT00003707
Title: A Phase I, Maximum Tolerated Dose (MTD) Trial to Determine the Safety and Pharmacokinetics of Chronic Oral Administration of Farnesyl Transferase Inhibitor R115777 in Combination With Gemcitabine in Subjects With Advanced Incurable Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066815; P30CA054174 (NIH); UTHSC-9785011335 (Other: UTHSCSA IRB); JRF-R115777-USA-4A (Other: Johnson and Johnson); SACI-IDD-98-03 (Other: San Antonio Cancer Institute); NCI-V98-1501 (Other: NCI)
Record Dates: First submitted 1999-11-01; First posted 2003-07-15 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Gemcitabine; tipifarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: tipifarnib

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase I trial to study the effectiveness of combining R115777 with gemcitabine in treating patients with advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and dose limiting toxicities of tipifarnib in combination with gemcitabine in patients with advanced cancer.
* Investigate potential pharmacokinetic interactions between tipifarnib and gemcitabine in these patients.
* Determine the efficacy of this regimen in patients with measurable or evaluable disease.
* Evaluate the quality of life of these patients.

OUTLINE: This is a dose-escalation study of tipifarnib.

Patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15 and oral tipifarnib every 12 hours beginning on day 2. Treatment continues every 4 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients each receive escalating doses of tipifarnib until the maximum tolerated dose (MTD) is reached. The MTD is defined as the dose at which fewer than one third of the patients experience dose limiting toxicity.

Quality of life is assessed before treatment, on day 22 of each course, and at the end of treatment.

PROJECTED ACCRUAL: A maximum of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically proven advanced cancer for which no curative therapy exists

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 9 g/dL

Hepatic:

* Bilirubin normal
* SGOT and SGPT no greater than 2 times upper limit of normal (ULN) (no greater than 5 times ULN if liver metastases present)

Renal:

* Creatinine normal

Other:

* Unassisted oral or enteral intake sufficient to maintain a reasonable state of nutrition
* No concurrent medical condition that is likely to interfere with study participation
* No active visual disturbances that require intervention beyond corrective lenses
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior bone marrow transplantation
* No concurrent immunotherapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No prior high dose chemotherapy with bone marrow or stem cell rescue
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormone therapy (except megestrol acetate)

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No prior radiotherapy to 25% or more of bone marrow
* No concurrent radiotherapy (except palliative radiotherapy within the first 28 days of the study)

Surgery:

* Not specified

Other:

* At least 30 days since prior investigational therapy
* No concurrent investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 1998-10; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric K. Rowinsky, MD, Study Chair — San Antonio Cancer Institute
Locations (1):
- San Antonio Cancer Institute, San Antonio, Texas, United States